Title: Randomized Clinical Trial of Hypovitaminosis D Treatment in the Neurocritical

Care Unit

IRB#: IRB\_00091541 IND#: 131398

**Date:** 8/30/17

# Randomized Clinical Trial of Hypovitaminosis D Treatment in the Neurocritical Care Unit

Michael Karsy, MD, PhD¹; Andrea Brock, MD, MSc¹; Ilyas Eli, MD¹; Jian Guan, MD¹; Aatman Shah, MD¹, Al-Wala Awad, MD¹, Sarah Menacho, MD¹; Min S Park, MD¹

<sup>1</sup>Department of Neurosurgery, Clinical Neurosciences Center, University of Utah, 175 North Medical Dr. East, Salt Lake City, UT 84132, USA

#### 1. Abstract

Vitamin D has been shown as an important marker of prognosis in a variety of clinical settings, including overall mortality, acute respiratory distress syndrome (ARDS), infection/sepsis, asthma, cardiovascular disease, diabetes, and pediatric/medical/surgical intensive care unit outcomes. Vitamin D not only plays a role in bone maintenance, but also a variety of extra-axial functions including immunedysregulation and systemic inflammation. In addition, a number of randomized clinical trials support the supplementation of vitamin D as improving outcome in critical care patients. While the evaluation of vitamin D levels remains a standard-of-care at our institution, the widespread use of vitamin D monitoring and impact on neurocritical care patients remains limited. Our recent prospective observational study of vitamin D levels in neurocritical patients showed that deficiency (<20ng/ml) was highly associated with prolonged hospital stay and increased in-hospital mortality for emergent patients. Moreover, a number of limitations arise from this study due to its observational nature. This study proposes a randomized, double-blinded, placebo-controlled, single center evaluation of vitamin D supplementation in the neurocritical care patient population (Table 1). Patients admitted to the neurocritical care unit for emergent cases and with vitamin D deficiency (<20ng/ml) will undergo vitamin D serum draw on admission and be randomized to receive cholecalciferol/vitamin D3 supplementation (540,000 IU once orally) or placebo with the primary measured outcome being hospital length-of-stay. Secondary outcomes will include length of hospital course, length of ICU course, complications, adverse events, discharge Glasgow Outcome Score, in-hospital and 30-day mortality, as well as quality-of-life. Power analysis estimates 198 patients will be needed for each subgroup to determine a 2 day difference in length-of-stay, and we plan to recruit 218 patients per treatment arm to account for dropout, which will take approximately 6-9 months to recruit. Interim analysis and safety monitoring will be performed. We hypothesize that vitamin D supplementation may make a significant impact on reducing morbidity and mortality in the neurocritical care population. The possibility of reducing hospital length of stay and mortality from a simple and cheap intervention such as vitamin D supplementation may be a useful adjuvant treatment in the neurocritical care population.

# 2. Background/Rationale

Hypovitaminosis D has a high prevalence among the general population, with some studies showing over half of the elderly population being affected (Chapuy 1997). Among critically ill patients, various studies have shown associations between hypovitaminosis D and multiple negative outcomes including mortality (De Haan 2014,

Rech 2014), ARDS (Dancer 2015), and infection (Flynn 2012). Vitamin D deficiency has also been shown to have impacts on various neurological diseases such as stroke (Yalbuzdag 2015, Chung 2015), and dementia (Littlejohns 2014). While the mechanism between vitamin D deficiency and these diseases is not entirely known, evidence suggest that vitamin D can affect vascular reactivity, inflammation, and the immune system (Carthy 1989, Vargas-Vasserot 2011) (Table S1, Figure S1-2).

Vitamin D has been shown to impact prognosis in a variety of retrospective and randomized clinical trials within an intensive care unit (ICU) environment (Amrein 2011). Despite these findings, there have been no studies examining the impact of hypovitaminosis D in specialized neurocritical care units (NCCU). Given the often significant differences in the management of patients in NCCU and more generalized intensive care units (Kurtz 2011) there is a need for further inquiries into the impact of low vitamin D levels in this specific environment. This study proposes a randomized, double-blinded, placebo-controlled, single center evaluation of vitamin D supplementation in the emergent NCCU patient population (Table 1). We have previously conducted a prospective, observational analysis of 823 NCCU patients and shown a significant reduction in hospital length-of-stay for all patients (7.14 vs. 5.97 days, p=0.0018) and for emergent cases (8.21 vs. 6.36 days, p=0.038), as well as reduced in-hospital mortality for emergent patients with non-deficient vitamin D levels (26/203 vs. 22/321, p=0.021). Nevertheless, these results remain limited in being observational studies without randomization or controls.

# 3. Study purposes and objectives

- 1. Evaluate the impact of vitamin D supplementation on the length-of-stay of emergent neurocritical care patients (primary outcome)
- 2. Evaluate the impact of vitamin D supplementation on in-hospital mortality, ICU length-of-stay, Glasgow Outcome Score on discharge, complications, and quality-of-life metrics (secondary outcome)
- 3. Evaluate the impact of vitamin D supplementation on Glasgow Outcome score and quality-of-life metrics at 3 and 6 months post-discharge (secondary outcome)

## 4. Methods

#### 4.1. Inclusion criteria

- Patients >18 years of age
- Patients admitted to the neurosurgery or neurology services
- Patients admitted to a critical care unit
- Informed consent
- Expected to stay in the ICU for 48 hours or more
- Vitamin D deficiency (<20ng/ml)

#### 4.2. Exclusion criteria

- Patients where a vitamin D level was not drawn within 48 hours of admission
- Patients not randomized within 48 hours of admission.
- Readmitted patients to the critical care unit
- Lack of informed consent

- Prior supplementation with vitamin D
- Severely impaired gastrointestinal function
- Other trial participation
- Pregnant or lactating women
- Hypercalcemia (total calcium of >10.6 mg/dL or ionized serum calcium of >5.4 mg/dL
- Tuberculosis history or clinical exam
- Sarcoidosis history or clinical exam
- Nephrolithiasis within the prior year
- Patients not deemed suitable for study participation (ie, psychiatric disease, living remotely from the clinic, or prisoner status)
- Pregnant or nursing women

## 4.3. General protocol

- 1. Patients will be identified through primary treatment teams, including the Departments of Neurosurgery and Neurology, and through screening of the electronic medical record for patients admitted to the NCCU at the University of Utah Health Sciences Center. Patients admitted for non-elective indications as outlined in the inclusion criteria will be enrolled. The full inclusion and exclusion criteria are listed in Table 1. We expect most patients to be admitted to the neurosurgery service and NCCU.
- 2. A Vitamin D level will be drawn on all non-electively admitted NCCU patients as part of our standard admission protocol.
- 3. Patients with a Vitamin D level <20ng/ml, defined as deficient, will be consented for the trial. Patients that do not consent for the trial will be studied retrospectively as part of our standard-of-care similarly to our previous prospective trial. Women between 18-45 years of age will undergo a serum or urine pregnancy test to rule out pregnancy prior to enrollment.</p>
- 4. Patients will be randomized 1:1 to receive Cholecalciferol (Vitamin D3, 540,000 IU once orally or by feeding) immediately or placebo by random number generator. Treatments will be blinded to the patient and physician care teams. Placebos will include similar tablets or liquid formulations that mimic the treatment drug but are indistinguishable.
- 5. A subsequent Vitamin D level will be drawn 3 days after drug administration or on date of discharge if sooner than 3 days to evaluate the adequacy of vitamin D repletion.
- 6. Primary outcomes will total hospital length-of-stay. Secondary outcomes will include in-hospital mortality, ICU length-of-stay, ICU complications (rates of sepsis/bacteremia, pneumonia, urinary tract infection), discharge Glasgow Outcome Score, medication adverse events, and quality-of-life metrics. Various patient demographic data will be acquired.
- 7. Subsequent 30-day mortality will be measured on standard clinical followup.

8. 1, 3 month and 6 month Glasgow Outcome Scores and quality-of-life metrics will be obtained. Physical therapy gait distance measurements as well as modified Rankin scale on discharge will be obtained.

## 4.4. Safety monitoring

There are minimal risks related to the patient. Vitamin D treatment is a relatively safe procedure in properly selected individuals. There may be additional discomforts including close monitored by the research team in order to monitor the study and collect data. The risk and side effects for Vitamin D administration are minimal and discussed further in the drug description. We have outlined a detailed data and safety monitoring plan.

We have previously shown Vitamin D administration in our prospective, observational study for patients with Vitamin D levels <10ng/ml to be safe and without any adverse effect at dosages of 50,000 IU Qweek of ergocalciferol/vitamin D2. The dosages used in this study are comparable to other studies evaluating Vitamin D efficacy and safety (Bacon 2009, Von Restorff 2009, Amrein 2011, Amrein 2014). There was no reported adverse event from ergocalciferol/vitamin D2 administration during our prospective, observational trial along with recent trials evaluating cholecalciferol/vitamin D3.

For patient safety, we will continue daily monitoring of CBC, BMP, Calcium, Phosphate, and neurological examinations as per standard practice in the neurocritical care unit. Should risks be identified, modification of the protocol will be proposed. And should the trial prove unsafe, we plan to notify the IRB and terminate the study. The study principal investigator and co-investigators will be responsible for oversight of patient safety. In addition, an independent safety and data review committee of licensed physicians will evaluate the study data on a quarterly basis. Quarterly safety and data monitoring reports will be discussed among the investigators and safety committee. The study will remain double-blinded except in the case of possible safety issues warranting unblinding.

Participants will be withdrawn from the study should they demonstrate >grade 3 Common Terminology Criteria for Adverse Events (CTCAE) suggesting Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated. In addition, patients will be withdrawn from the study should they show other signs/symptoms of vitamin D toxicity including, hypercalcemia, anorexia, nausea, vomiting, as well as polyuria, polydipsia, weakness, nervousness, pruritus, laboratory studies suggesting renal injury or failure (proteinuria, urinary casts, azotemia, metastatic renal calcifications). A checklist will be used to monitor patients. These findings can be uncovered by routine neurological and laboratory exams as per the ICU standard. Should adverse events be identified at higher or clustered rates than expected statistically, the trial will be modified or terminated.

#### 4.5. Informed consent

The goals of the study, including potential benefit and minimal risk, will be discussed. Patients will be told that not participating in the study will not affect their hospital care. We will provide patients with a copy of the informed consent containing contact information for the investigators. In addition, we will inform the critical care staff,

including nursing and administration, regarding the study so patients can find the appropriate research staff should they have questions. All interim and data safety analysis when analyzed will be immediately conveyed to all study participants in the event of potential adverse events or risks.

In some cases a legally authorized representative (LAR) will be used for informed consent of the patient. Many of the emergent patients admitted to the NCCU will not have the capacity for an informed consent. LARs may include spouses or patient children, as well as authorized legal healthcare proxies, depending on policies for informed consent at the University of Utah Health Sciences Center. As with studies of Vitamin D in other critical care settings, patient consent through a proxy may be possible. We will include a LAR signature block at the end of the consent document.

Phone consents will be allowed as part of the trial to ensure timely consent. Similar, to surgical or procedural consents, phone consents will involve discussion with a LAR and informed consent will be documented by the study investigator as well as a witness, usually the patient's nurse. Phone consents will be performed when the patient is incapacitated and family is unable to reach the hospital to sign the paper consent.

# 4.6. Privacy protection

Information about each participant, including the results of tests, will be confidential. Each participant will be assigned a study number and we will not use the participant's name in our study records. Paper records will be kept in a locked file cabinet in a secure room. Computerized records will be kept in a locked room on password-protected computers. The participant's name will not be used in any published reports.

#### 4.7. Facilities and staff

The principal investigator and co-investigators are all licensed physicians within the department of neurosurgery with experience in both basic and clinical science research. All investigators have had prior database research experience, including IRB submission as well as data acquisition and analysis. The faculty advisor, is a licensed physician as well as a board-certified neurosurgeon and Assistant Professor at the University of Utah, has also reviewed the protocol and will be involved in patient safety monitoring as well as quality control. He has been involved in our prior prospective, observational study on Vitamin D status of neurocritical care patients. The project will be discussed by meetings and by email as necessary to discuss results, patient safety issues, and data quality. All investigators are already trained in research methodology, have completed CITI certification, receive annual training on research bioethics through the Department of Neurosurgery, and have been trained on aspects of informed consent.

The research will be primarily performed at the University of Utah Hospital. Some data analysis may be performed on computers within the Neurosciences Center at the University. The NCCU at the University Hospital will be the predominant facility used for research activity. Other ICUs will be used if neurosurgery or neurology patients are admitted. All information related to be data will be kept in a HIPAA-compliant database or locked cabinet units only accessed by the principal investigator. The University of Utah Neurocritical Care Unit (NCCU) NCCU is a 23-bed intensive care unit which

specializes in the treatment of patients with critical neurological illness, such as stroke, intracranial hemorrhage, status epilepticus, traumatic brain injury, and meningitis. The NCCU is the region's largest and most technologically advanced critical care unit and the catchment are for the NCCU comprises 20% of the geographical area of the continental United States. Nurses specially trained in caring for neurological patients who require intensive care staff the NCCU in conjunction with 5 neurointensivists and a multidisciplinary team of neurologists and neurosurgeons.

# 4.8. Selection of therapeutic agent

Patients will be supplemented with cholecalciferol (vitamin D3) or placebo. Two major vitamin D compounds exist in humans, ergocalciiferol (vitamin D2) and cholecalciferol (vitamin D3) and recent guidelines suggest that either vitamin D2 or vitamin D3 can be supplemented in patients with hypovitaminosis D (Holick 2011). One study evaluating short-term supplementation with vitamin D2 in an critical care setting demonstrate that only 26% of patients receiving 50,000 IU three times per week achieved normal vitamin D levels (Dickerson 2015). Critically ill patients have been suggested to have a blunted response to vitamin D supplementation. Nonetheless, a number of randomized trials have shown the ability of high dose vitamin D3 to adequate replete critically ill patients with minimal toxicity, mostly mild hypercalcemia (Quraishi 2015, Nair 2015, Amrein 2011, Amrein 2014). Intramuscular (200,000 IU) or oral (540,000 IU) have been shown to adequately replete vitamin D levels in the majority of patients by 2-7 days after treatment. For this reason we have chosen to supplement with cholecalciferol (540,000 IU) orally).

## 4.9. Power analysis and statistical plan

A variety of variables will be collected on patients (Table 2). We estimated various sample sizes based on our preliminary, prospective, observational trial. Using length-of-stay as a primary outcome, previously we detected a significant decrease in patients with sufficient vitamin D levels (>20ng/ml) (8.21 vs. 6.36 days, p=0.002). Using an effect size of 2, alpha of 0.05, 1:1 case/control sampling, we estimate 198 patients will be required per group for this study. We plan to recruit patients to account for a 10% dropout resulting in 218 patients per group, total 436. We also performed power calculations using various other outcomes including, in-hospital mortality, as well as evaluation of both emergent and non-emergent patients. Based on a 6-month timeframe needed to enroll 512 patients in our prospective, observational trial, we estimate the trial would take 12 months for enrollment and randomization in the proposed trial. The primary outcome (length-of-stay) will be measured by T-test as well as multivariate regression to adjust for potential confounders using SPSS (IBM, Armonk, NY). Secondary outcomes will be evaluated by a variety of statistical methods.

### 4.10. Funding source

Planned sources of funding for this study are from internal departmental grants without potential for conflicts-of-interest. No submission for additional funding sources is planned at this time.

# 5. Anticipated results and potential public health impact

The potential benefit of this study would include knowledge about the success of vitamin D supplementation on various critical care outcomes. While they may not directly apply to a patient, they can be useful to additional critical care patients admitted an ICU in the future. The societal benefit will include reduced patient morbidity and mortality, as well as shorter hospital stays and therefore reduced ICU expenditure. Vitamin D is a relatively cost-effective medication that is well-tolerated. Its potential impact to reduce hospital stays, by even 1 day would play a significant role in reducing patient cost, disease morbidity, and risk from hospitalization. Future research directions can involve a multi-center randomized clinical trial to validate the effect of vitamin D in the neurocritical care patient as well as further molecular studies evaluating the non-skeletal effects of vitamin D. Additional, studies on vitamin D as a biomarker and effects on a cellular level can also be forthcoming if a potential benefit is identified clinically. Identification of the molecular mechanisms by which vitamin D may alter disease pathology may serve as a method for the development of additional treatments.

### 6. Protocol amendments

- 6.1. 1/10/17, Addition of phone consents as well as two study co-investigators, Aatman Shah, MD and Al-Wala Awad, MD was performed. Repeat vitamin D levels at 3 days following administration of study drug or placebo was modified from prior planned repeat vitamin D at 7 days.
- 6.2. 8/6/17, Addition of physical therapy assessment and modified Rankin scale as secondary outcomes of the study. Change of study faculty sponsor from Dr. Min S. Park to Dr. Sarah T. Menacho as Dr. Park is leaving the University of Utah.

| Table 1: Summary | of Study Characteristics |
|---|---|
| Title | Randomized Clinical Trial of Hypovitaminosis D Treatment in |
| | the Neurocritical Care Unit |
| Methodology | Randomized, double-blinded, placebo-controlled clinical trial |
| Study Duration | 1-1.5 years (12 months recruitment, 3-6 month analysis) |
| Study Center(s) | University of Utah Health Sciences Center |
| Objectives | Evaluate the impact of vitamin D supplementation on the |
| | length-of-stay of emergent neurocritical care patients (primary |
| | outcome) |
| | 2. Evaluate the impact of vitamin D supplementation on in- |
| | hospital mortality, ICU length-of-stay, Glasgow Outcome Score |
| | on discharge, complications, and quality-of-life metrics |
| | (secondary outcome) |
| Primary Aims | Length-of-stay |
| Secondary Aims | ICU length-of stay, in-hospital mortality, 30-day mortality, ICU |
| | complications (sepsis, pneumonia, urinary tract infection), |
| | Glasgow Outcome Score, medication adverse events, modified |
| | Rankin Scale, physical therapy assessments |
| Number of | 218 per treatment arm, total 436 |
| Subjects | |
| Intervention | Vitamin D3 540,000 IU oral vs. placebo |
| Diagnosis and | Patients >18 years of age |
| Main Inclusion | Patients admitted to the neurosurgery or neurology services |
| Criteria | Patients admitted to a critical care unit |
| | Informed consent |
| | Expected to stay in the ICU for 48 hours or more |
| Exclusion criteria | Vitamin D deficiency (<20ng/ml) Patients where a vitamin D level was not drawn within 48 hours of |
| Exclusion chilena | admission |
| | Patients not randomized within 48 hours of admission |
| | Readmitted patients to the critical care unit |
| | Lack of informed consent |
| | Prior supplementation with vitamin D |
| | Severely impaired gastrointestinal function |
| | Other trial participation |
| | Pregnant or lactating women |
| | Hypercalcemia (total calcium of >10.6 mg/dL or ionized serum |
| | calcium of >5.4 mg/dL |
| | Tuberculosis history on clinical exam |
| | Sarcoidosis history on clinical exam |
| | Nephrolithiasis within the prior year |
| | Patients not deemed suitable for study participation (ie, psychiatric |
| | disease, living remotely from the clinic, or prisoner status) |
| | Pregnant or nursing women |
| Data and safety | Monthly review of data entry |

| monitoring | Quarterly independent review of data safety metrics |
|---|---|
| | Daily review of patient neurological exam, and laboratory values |
| | (CBC, BMP, calcium, phosphate) |
| | Interim 6-month data analysis |
| Statistical | T-test (parametric), Chi-square (non-parametric), univariate |
| Methodology | regression, multivariate linear regression, logistic regression, |
| | Kaplan-Meier survival, Cox proportional hazards modeling, interim |
| | analysis |
| | SPSS (IBM, Armonk, NY) |

# Table 2: Demographic, Clinical, and Safety Variables

# **Demographic Variables**

- Name
- Medical record number
- Date of birth
- Gender
- Diagnosis
- Ethnicity/race

#### **Clinical Variables**

- Date of admission to NCCU
- Disease category (tumors, trauma, vascular, other)
- Disease severity: Glasgow Coma Scale, Simplified Acute Physiology Score II
- Medical comorbidities: diabetes, hypertension, heart disease, cancer history
- Any surgeries during hospitalization
- Randomization vitamin D or placebo
- Vitamin D level on admission
- Date vitamin D level
- Vitamin D level 3 days post treatment
- Date vitamin D level 3 days post treatment
- Date ICU discharge
- Date hospital discharge
- Date deceased
- Glasgow Outcome Score on discharge
- EQ-5D on discharge
- Discharge disposition
- Hospital complications (specifically: deep vein thrombosis, bacteremia, urinary tract infection, pneumonia, readmission to NCCU)
- Glasgow Outcome Score at 3 and 6 months
- EQ-5D at 1, 3 and 6 months
- Physical therapy assessments at discharge
- Modified Rankin Scale on discharge

### Safety Monitoring

- Common Terminology Criteria for Adverse Events (CTAE) V4.0
- Daily ICU laboratory studies (CBC, BMP, calcium, phosphate)
- Daily neurological exam
- · Quarterly independent review of safety and data
- Monitoring of adverse events

| Table S1: Clinical Studies Evaluating Vitamin D in a Critical Care Environment | | | |
|---|---|---|---|
| Reference | Study type | Participants/ | Summary |
| | | groups | |
| Van den<br>Berghe<br>2003 | RCT | 22<br>200 IU vs. 500IU | Minimal change in serum markers |
| Ostermann<br>2007 | Retrospective cohort | 100<br>Normal vs.<br>insufficient vs.<br>deficient | Hospital-free days were significantly different between patients with deficiency and sufficiency No significant relationship between 25(OH)D concentrations and mortality |
| Lucidarme<br>2010 | Retrospective cohort | 100<br>Normal vs.<br>insufficient vs.<br>deficient vs.<br>undetectable | 28-day mortality was significantly different between the four groups No significant association between 25(OH)D concentrations and length of ICU stay. 79% of patients had low 25(OH)D concentrations |
| Mata-<br>Granados<br>2010 | RCT | 33<br>Placebo vs. 60,000<br>IU PO, vs. 2mcg IV<br>vit D3 | 97% of critically ill patients were vitamin D deficient. Group B (60,000 IU) showed a statistically significant increase in 25(OH)D concentrations. |
| Cecchi 2011 | Retrospective cohort | 170<br>Severe sepsis vs.<br>non-septic trauma | 28-day mortality was not statically different between the two groups with rates of 27.9% in severe septic patients and 11.1% in trauma patients |
| Braun 2011 | Retrospective cohort | 2,399<br>Normal vs.<br>insufficient vs.<br>deficient | Preadmission 25(OH)D deficiency is associated with mortality Adjusted 30-day morality odds ratio was 1.00, 1.36, and 1.69, respectively |
| Amrein 2011 | RCT | 25<br>Placebo vs.<br>540,000 IU enteral | The mean serum 25(OH)D increased in the treatment group 25 ng/mL. Deficiency was corrected in 2 days with |
| Venkatram<br>2011 | Retrospective cohort | 437<br>Normal vs.<br>insufficient vs. | Higher hospital mortality for patients with vitamin D deficiency but not insufficiency |

| | | deficient | |
|---|---|---|---|
| Braun<br>2012a | Retrospective cohort | 1,325<br>Normal vs.<br>insufficient vs.<br>deficient | Adjusted 30-day mortality odds ratio was 1.00, 1.35, and 1.94 b respectively |
| Braun<br>2012b | Retrospective cohort | 2,075<br>Normal vs.<br>insufficient vs.<br>deficient | Adjusted 30-day mortality odds ratio was 1.00, 1.41, and 1.61, respectively Preadmission 25(OH)D deficiency is significantly associated with acute kidney injury |
| Arnson 2012 | Prospective cohort | 130<br>Normal vs.<br>insufficient | Mortality was lower for vitamin D deficient patients (15±12.4 days vs. 24.2 ± 16.5 days) Vitamin D levels correlated with WBC count |
| Flynn 2012 | Prospective cohort | 66<br>Normal vs. deficient | Longer length of stay, infection rates and rates of sepsis in patients with vitamin D deficiency |
| Higgins<br>2012 | Prospective cohort | 196<br>Normal vs. deficient<br>vs. insufficient | Vitamin D levels decreased 3 days after admission and remained through 10 days Higher vitamin D levels were associated with shorter time to ICU discharge (HR 2.11) Vitamin D not associated with mortality or infection rate |
| Nair 2012 | Prospective cohort | 100<br>Normal vs. deficient<br>vs. insufficient | Vitamin D deficiency associated with fewer hospital-free days. Secondary hyperparathyroidism was highly prevalent in the critically ill population |
| Remmelts<br>2012 | Prospective cohort | 272<br>Normal vs. deficient<br>vs. insufficient | Vitamin D deficiency associated with increased risk of ICU admission and 30-day mortality in patients with community-acquired pneumonia |
| Nair 2013 | Retrospective cohort, RCT | 196 Normal vs. insufficient vs. deficient Placebo vs. low (200IU) vs. high (500IU) supplement | Mean time-to-alive at ICU discharge was 5.9 ± 5.4, 6.8 ± 6.0, and 10.6 ±8.4 respectively 25(OH)D insufficiency was not associated with mortality 25(OH)D levels were higher in the high dose group on days 2, 6, and 7. Doses studied did not |

| | | | normalize 25(OH)D serum |
|---|---|---|---|
| | | | concentrations |
| Aygencel<br>2013 | Prospective cohort | 201 | Increased mortality in vitamin D deficient (<20ng/mL) patients (43 vs. 26%) Increase rates of severe acute disease, worsened laboratory studies on admission, morbidity and exposure to invasive therapy in deficient patients. |
| Su 2013 | Prospective cohort | 206 (105 ICU)<br>Normal vs. ICU<br>sepsis | Lower vitamin D seen in patients with ICU sepsis compared to normal patients No difference in mortality with vitamin D levels |
| Amrein 2014 | RCT | 475, (patients with deficiency ≤20 ng/ml) Placebo vs. 540,000 IU x1, monthly 90,000 IU for 5 month | No difference in mean hospital stay (19.3 vs. 20.1), hospital mortality (35.3% vs. 28.3%), 6-month mortality (42.9% vs. 35.0%) Severe vitamin D subgroup (n=200) showed no difference in hospital stay (19 vs 20.1 days) and 6-month mortality (50% vs. 34.7%) Severe vitamin D subgroup showed significantly lower hospital mortality (46.1% vs. 28.6%, p=0.04), |
| Moromizato<br>2014 | Retrospective<br>cohort, two-<br>center | 3,386<br>Normal vs.<br>insufficiency vs.<br>deficiency | Preadmission vitamin D deficiency was predictive for risk of sepsis including after adjustement for other variables 90-day mortality was 1.6x higher in patients with preadmission vitamin D insufficiency and deficiency (HR. 1.63) |
| Dickerson<br>2015 | Retrospective cohort | 65<br>50,000 IU qweek,<br>Blweek, Tlweek for<br>4 weeks | Normal vitamin D levels achieved in 6%, 11% and 26% of patients |
| Brook 2015 | Retrospective cohort | 300<br>Normal vs. deficient | Vitamin D levels showed an inverse correlation with non-home discharge destination |
| Nair 2015 | RCT | 50<br>150,000 IU vs. | 65% vs. 67% of patients normalized vitamin D levels by 7 |

| | | 300,000 IU vitamin<br>D3 IM | days 80% vs. 83% of patients normalized vitamin D levels by 14 days Secondary hyperparathyroidism manifest in 25% of patients |
|---|---|---|---|
| Alizadeh<br>2015 | Retrospective cohort | 70<br>Normal vs. deficient | Longer length of stay (7.8 vs. 4.05 days) with deficient patients but no difference in hospital mortality |
| Quraishi<br>2015 | RCT | 30<br>Placebo vs.<br>200,000 IU<br>cholecalciferol vs.<br>400,000 IU<br>cholecalciferol | Plasma levels of vitamin D peaked on day 5 of treatment CRP levels did not differ between groups |
| Verceles<br>2015 | Retrospective cohort | 183<br>Normal vs. deficient | Deficiency was common (61% patients) and not associated with days to wean from ventillation |

| | Vit D | - Vit D+ | • | Risk Ratio | Risk Ratio |
|---|---|---|---|---|---|
| Study | Total | Total | Weight | IV, Random, 95% CI | IV, Random, 95% CI |
| Braun, 2011 [3] | 637 | 844 | 41.0% | 1.69 [1.28, 2.23] | ■ |
| Braun, 2012 [5] | 668 | 185 | 27.3% | 1.85 [1.15, 2.98] | - <b>-</b> - |
| Higgins, 2012 [23] | 50 | 37 | 9.9% | 0.68 [0.25, 1.84] | -+ |
| Lucidarme, 2010 [16] | 35 | 28 | 8.1% | 0.45 [0.14, 1.40] | <del></del> + |
| Nair, 2012 [27] | 24 | 21 | 5.4% | 1.42 [0.34, 5.91] | <del></del> |
| Remmelts, 2012 [28] | 143 | 50 | 4.8% | 2.40 [0.52, 11.03] | + |
| Su, 2013 [29] | 129 | 6 | 3.5% | 1.44 [0.23, 8.86] | <del></del> |
| Total (95% CI) | 1686 | 1171 | 100.0% | 1.42 [1.00, 2.02] | <b>*</b> |
| Heterogeneity: Tau <sup>2</sup> = 0.06; Chi <sup>2</sup> = 8.45 | , df = 6 (P = 0.21) | ); I <sup>2</sup> = 2 | 9% | H | |
| Test for overall effect: Z = 1.98 (P = 0.0 | 5) | | | | 0.01 0.1 1 10 100<br>[Vit D+] [Vit D-] |

Figure S1: Forest plot of 30-day mortality in studies with univariate analysis of vitamin D sufficiency vs. deficiency. Adapted from de Haan et al. 2014.

| | Vit D- | Vit D+ | | Risk Ratio | Risk Ratio |
|---|---|---|---|---|---|
| Study | Total | Total | Weight | IV, Random, 95% CI | IV, Random, 95% CI |
| Amrein, 2014 [25] | 349 | 89 | 20.6% | 1.97 [1.31, 2.97] | -1- |
| Aygencel, 2013 [24] | 139 | 62 | 16.0% | 1.67 [1.05, 2.66] | - |
| Braun, 2011 [3] | 637 | 844 | 44.4% | 1.77 [1.34, 2.34] | - ■ |
| Braun, 2012 [5] | 668 | 185 | 13.5% | 1.92 [1.16, 3.18] | - |
| Flynn, 2012 [22] | 49 | 17 | 1.0% | 0.49 [0.07, 3.21] | <del></del> |
| Matthews, 2012 [30] | 138 | 21 | 0.4% | 6.19 [0.36, 106.88] | <del></del> |
| Nair, 2012 [27] | 24 | 21 | 3.2% | 1.05 [0.37, 2.95] | |
| Venkatram, 2011 [4] | 340 | 23 | 0.8% | 6.99 [0.93, 52.68] | - |
| Total (95% CI) | 2344 | 1262 | 100.0% | 1.79 [1.49, 2.16] | • |
| Heterogeneity: Tau <sup>2</sup> = 0.00; Chi <sup>2</sup> = 5.71, df = 7 ( | P = 0.57) | ; I <sup>2</sup> = 0% | , | <b>⊢</b> | <del></del> |
| Test for overall effect: Z = 6.16 (P < 0.001) | , | | | 0.0 | 1 0.1 1 10 100<br>[Vit D+] [Vit D-] |

Figure S2: Forest plot of in hospital mortality in studies with univariate analysis of vitamin D sufficiency vs. deficiency. Adapted from de Haan et al. 2014.

#### 7. Reference

Alizadeh N, Khalili H, Mohammadi M, Abdollahi A. Serum Vitamin D levels at admission predict the length of intensive care unit stay but not in-hospital mortality of critically ill surgical patients. J Res Pharm Pract. 2015 Oct-Dec;4(4):193-8

Amrein, K.; Sourij, H.; Wagner, G.; Holl, A.; Pieber, T.R.; Smolle, K.H.; Stojakovic, T.; Schnedl1, C.; Dobnig, H. Short-term effects of high-dose oral vitamin D3 in critically ill vitamin D deficient patients: a randomized, double-blind, placebo-controlled pilot study. Crit. Care 2011.

Amrein K, Schnedl C, Holl A, Riedl R, Christopher KB, Pachler C, Urbanic Purkart T, Waltensdorfer A, Münch A, Warnkross H, Stojakovic T, Bisping E, Toller W, Smolle KH, Berghold A, Pieber TR, Dobnig H. Effect of high-dose vitamin D3 on hospital length of stay in critically ill patients with vitamin D deficiency: the VITdAL-ICU randomized clinical trial.

JAMA. 2014 Oct 15;312(15):1520-30

Arnson Y, Gringauz I, Itzhaky D, Amital H: Vitamin D deficiency is associated with poor outcomes and increased mortality in severely ill patients. QJM 2012, 105:633 639.

Aygencel G, Turkoglu M, Tuncel AF, Candir BA, Bildaci YD, Pasaoglu H: Is vitamin D insufficiency associated with mortality of critically ill patients? Crit Care Res Pract 2013, 2013:856747.

Bacon CJ,Gamble GD, Horne AM, Scott MA, Reid IR. High-dose oral vitamin D3 supplementation in the elderly. *Osteoporos Int*. 2009;20(8):1407-1415.

Braun, A.; Chang, D.; Mahadevappa, K.; Christopher, K.B. Association of low serum 25-hydroxyvitamin D levels and mortality in the critically ill. Crit. Care Med. 2011, 39, 671–677.

Braun, A.B.; Gibbons, F.K.; Litonjua, A.A.; Giovannucci, E.; Christopher, K.B. Low serum

25-hydroxyvitamin D at critical care initiation is associated with increased mortality. Crit. Care Med. 2012, 40, 63–72.

Braun, A.B.; Litonjua, A.A.; Moromizato, T.; Gibbons, F.K.; Giovannucci, E.; Christopher, K.B.

Association of low serum 25-hydroxyvitamin D levels and acute kidney injury in the critically ill. Crit. Care Med. 2012, 40, 3170–3179

Brook K, Camargo C.A., Christopher K.B., Quraishi S.A.; Admission vitamin D status is associated with discharge destination in critically ill surgical patients. Ann Intensive Care. 2015 Dec;5(1):23

Carthy EP, Yamashita W, Hsu A, Ooi BS. 1,25-dihydroxyvitamin D3 and rat vascular smooth muscle cell growth. Hypertension. 1989;13:954-9.

Cayir A, Turan MI, Ozkan O, Cayir Y. Vitamin D levels in children diagnosed with acute otitis media. J Pak Med Assoc. 2014;64(11):1274-7.

Cecchi, A.; Bonizzoli, M.; Douar, S.; Mangini, M.; Paladini, S.; Gazzini, B.; Degl'Innocenti, S.;

Linden, M.; Zagli, G.; Peris, A. Vitamin D deficiency in septic patients at ICU admission is not a mortality predictor. Minerva Anestesiol. 2011, 77, 1184–1189, (in Italian).

Chapuy MC, Preziosi P, Maamer M, Arnaud S, Galan P, Hercberg S, meunier PJ. Prevalence of vitamin D insufficiency in an adult normal population. Osteoporos Int. 1997;7(5):439-43.

Chung PW, Park KY, Kim JM, Shin DW, Park MS, Chung YJ, Ha SY, Ahn SW, Shin HW, Kim YB, Moon HS. 25-hydroxyvitamin D status is associated with chronic cerebral small vessel disease. Stroke. 2015;46(1):248-51.

De Haan K, Groeneveld AB, de Geus HR, Egal M, Struijs A. Vitamin D deficiency as a risk factor for infection, sepsis and mortality in the critically ill: systematic review and meta-analysis

Critical Care 2014, 18:660

Dickerson RN, Berry SC, Ziebarth JD, Swanson JM, Maish GO, Minard G, Brown RO. Dose-response effect of ergocalciferol therapy on serum 25-hydroxyvitamin D concentration during critical illness. Nutrition. 2015 Oct;31(10):1219-23

Flynn L, Zimmerman LH, McNorton K, Dolman M, Tyburski J, Baylor A, Wilson R, Dolman H: Effects of vitamin D deficiency in critically ill surgical patients. Am J Surg 2012, 203:379 382

Giovannucci E, Liu Y, Rimm EB, Hollis BW, Fuchs CS, Stampfer MJ, Willett WC. Prospective study of predictors of vitamin D status and cancer incidence and mortality in men. J Natl Cancer Inst. 2006;98(7):451-9.

Dancer RC, Parekh D, Lax S, D'Souza V, Zheng S, Bassford CR, Park D, Bartis DG, Mahida R,

De Haan K, Groeneveld AB, de Geus HR, Egal M, Struijs A. Vitamin D deficiency as a risk factor for infection, sepsis and mortality in the critically ill: systemic review and meta-analysis. Crit Care. 2014;18(6):660.

Dickerson RN, Berry SC, Ziebarth JD, Swanson JM, Maish 3rd GO, Minard G, et al. Dose-response effect of ergocalciferol therapy on serum 25-hydroxyvitamin D concentration during critical illness. Nutrition. 2015;31(10):1219–23.

Flynn L, Zimmerman LH, McNorton K, Dolman M, Tyburski J, Baylor A, Wilson R, Dolman H. Effects of vitamin D deficiency in critically ill surgical patients. Am J Surg. 2012;203(3):379-82.

Higgins DM, Wischmeyer PE, Queensland KM, Sillau SH, Sufit AJ, Heyland DK: Relationship of vitamin D deficiency to clinical outcomes in critically ill patients. J Parenter Enter Nutr 2012, 36:713 720.

Khoo AL, Chai LY, Koenen HJ, Kullberg BJ, Joosten I, van der Ven AJ, Netea MG. 1,25-dihydroxyvitamin D3 modulates cytokine production induced by candida albicans: impact of seasonal variation of immune responses. J Infect Dis. 2011;203:122-130.

Kurtz P, Fitts V, Sumer Z, Jalon H, Cooke J, Kvetan V, Mayer SA. How does care differ for neurological patients admitted to a neurocritical care unit versus a general ICU. Neurocrit Care. 2011;15(3):477-80.

Leaf DE, Raed A, Donnino MW, Ginde AA, Waikar SS. Randomized controlled trial of calcitriol in severe sepsis. Am J Respir Crit Care Med. 2014;190(5):533–41.

Littlejohns TJ, Henley WE, Lang IA, Annweiler C, Beauchet O, Chaves PH, Fried L, Kestenbaum BR, Kuller LH, Langa KM, Lopez OL, Kos K, Soni M, Llewellyn DJ. Vitamin D and the risk of dementia and Alzheimer's disease. Neurology. 2014;83(10):920-8.

Lucidarme, O.; Messai, E.; Mazzoni, T.; Arcade, M.; du Cheyron, D. Incidence and risk factors of vitamin D deficiency in critically ill patients: results from a prospective observational study. Intensive Care Med. 2010, 36, 1609–1611.

Mata-Granados, J.M.; Vargas-Vasserot, J.; Ferreiro-Vera, C.; de Castro, L.; Pavón, R.G.;

Gómez, J.M.Q. Evaluation of vitamin D endocrine system (VDES) status and response to

treatment of patients in inten—sive care units (ICUs) using an on-line SPE-LC-MS/MS method. J. Steroid Biochem. Mol. Biol. 2010, 121, 452–455.

Moromizato T, Litonjua AA, Braun AB, Gibbons FK, Giovannucci E, Christopher KB: Association of low serum 25-hydroxyvitamin D levels and sepsis in the critically ill. Crit Care Med 2014, 42:97 107.

Nair P, Lee P, Reynolds C, Nguyen N.D., Myburgh, J., Eisman J.A., Center J.R. Significant perturbation of vitamin D-parathyroid-calcium axis and adverse clinical outcomes in critically ill patients. Intensive Care Med. 2013, 39, 267–274.

Nair P, Venketash B, Lee P, Kerr S, Hoechter D.J., Dimeski G, Grice J, Myburgh J, Center JR. A Randomized Study of a Single Dose of Intramuscular Cholecalciferol in Critically III Adults. Crit Care Med. 2015 Nov;43(11):2313-20.

Ostermann, M.; Chang, R.W. Acute kidney injury in the intensive care unit according to RIFLE. Crit. Care Med. 2007, 35, 1837–1843.

Quraishi S.A, De Pascale G, Needleman J.S., Nakazawa H, Kaneki M, Bajwa E.K., Camargo C.A, Bhan I. Effect of Cholecalciferol Supplementation on Vitamin D Status and Cathelicidin Levels in Sepsis: A Randomized, Placebo-Controlled Trial. Crit Care Med. 2015 Sep;43(9):1928-37.

Rech MA, Hunsaker T, Rodriguez J. Deficiency in 25-hydroxyvitamin D and 30-day mortality in patients with severe sepsis and septic shock. Am J Crit Care. 2014;23(5):e72-9.

Rousseau AF, Foidart-Desalle M, Ledoux D, Remy C, Croisier JL, Damas P, et al. Effects of cholecalciferol supplementation and op-timized calcium intakes on vitamin D status, muscle strength and bone health: a one-year pilot randomized controlled trial in adults with severe burns. Burns. 2015;41(2):317–25.

Su LX, Jiang ZX, Cao LC, Xiao K, Song JP, Li H, Zhang X, Yan P, Feng D, Liu CT, Li X, Xie LX: Significance of low serum vitamin D for infection risk, disease severity and mortality in critically ill patients. Chin Med J (Engl) 2013, 126:2725 2730.

Turner AM, Sapey E, Wei W, Naidu B, Stewart PM, Fraser WD, Christopher KB, Cooper MS, Gao F, Sansom DM, Martineau AR, Perkins GD, Thickett DR. Vitamin D deficiency contributes directly to the acute respiratory distress syndrome (ARDS). Thorax. 2015;70&7):617-24.

Van den Berghe G, Van Roosbroeck D, Vanhove P, Wouters PJ, De Pourcq L, Bouillon R. Bone turnover in prolonged critical illness: effect of vitamin D. J Clin Endocrinol Metab. 2003;88(10):4623–32.

Vargas-Vasserot J, Mata-Granados JM, Luque De Castro M, Guerrero Pavon R, Quesada Gomez J. 25-hydroxyvitamin D3 treatment normalizes the vitamin D status and the innate immune response mediated by cathelicidin in critically ill patients. Bone. 2011;48-S146-147.

Verceles A.C., Weiler B, Koldobskiy D, Goldberg A.P, Netzer G, Sorkin J.D. Association Between Vitamin D Status and Weaning From Prolonged Mechanical Ventilation in Survivors of Critical Illness. Respir Care. 2015 Jul;60(7):1033-9

Venkatram S, Chilimuri S, Adrish M, Salako A, Patel M, Diaz-Fuentes G. Vitamin D deficiency is associated with mortality in the medical intensive care unit. Crit Care. 2011;15(6):R292.

Von Restorff C, Bischoff-Ferrari HA, Theiler R. High-dose oral vitamin D3 supplementation in rheumatology patients with severe vitamin D3 deficiency. *Bone*.

2009;45(4):747-749.

Yalbuzdag SA, Sarifakioglu B, Afsar SI, Celik C, Can A, Yegin T, Senturk B, Guzelant AY. Is 25(OH)D associated with cognitive impairment and functional improvement in stroke? A retrospective clinical study. J Stroke Cerebrovasc Dis. 2015;24(7):1479-86.